CLINICAL TRIAL: NCT04831151
Title: The Effect of Two Combined Oral Contraceptives Containing Cyproterone Acetate or Drospirenone on Blood Metabolomics in Women With Polycystic Ovary Syndrome
Brief Title: The Effect of Polycystic Ovary Syndrome Treatment on Metabolomics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Senem Arda Düz, Assistant professor, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/28
Record Dates: First submitted 2021-03-28; First posted 2021-04-05 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Polycystic Ovary Syndrome
Keywords: hirsutism; combined oral contraceptives; amenorrhea
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hirsutism; Amenorrhea | interventions — drospirenone and ethinyl estradiol combination; Cyproterone acetate, ethinyl estradiol drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drospirenone group: 0,03 mg ethinylestradiol + 3 mg drospirenone (Active Comparator): generic name:yasmin dosage form:oral dosage: 0,03 mg ethinylestradiol + 3 mg drospirenone frequency: once a day duration: 3 months
  Interventions: Drug: Yasmin
- cyproterone acetate group: 0,035 mg ethinylestradiol + 2 mg cyproterone acetate (Active Comparator): generic name:diane 35 dosage form:oral dosage: 0,035 mg ethinylestradiol + 2 mg cyproterone acetate frequency: once a day duration: 3 months
  Interventions: Drug: Diane-35

INTERVENTIONS:
Drug: Yasmin — Yasmin: 0,03 mg ethinylestradiol + 3 mg drospirenone
  Arms: Drospirenone group: 0,03 mg ethinylestradiol + 3 mg drospirenone
Drug: Diane-35 — Diane 35: 0,035 mg ethinylestradiol + 2 mg cyproterone acetate
  Arms: cyproterone acetate group: 0,035 mg ethinylestradiol + 2 mg cyproterone acetate

SUMMARY:
The aim of this study is to determine the effect of the treatment of polycystic ovary syndrome with two different oral contraceptives that contain cyproterone acetate and drospirenone

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS), is the most common endocrinological disorder that affects the reproductive aged women. In addition to causing problems such as menstrual irregularity, hirsutism, acne, it is also an important health problem that can cause infertility, insulin resistance, impaired glucose metabolism, diabetes, high blood pressure, heart disease, dyslipidemia in advanced ages. Diagnostic criteria also vary widely in these patients. These patients are often overweight or obese, and abdominal adiposity is common in these patients. The patients also suffer from insulin resistance and hyperinsulinemia in this syndrome. All of this is probably the result of a vicious cycle that starts in the antenatal period. Combined oral contraceptives (COCs), are the first-choice treatment option for many patients by improving both menstrual irregularity, hyperandrogenism, and insulin resistance through sex hormone binding globulin (SHBG). They reduce the risk of endometrial hyperplasia and endometrial cancer by providing regular menstruation.

Nowadays, the use of metabolomics is increasing in understanding the pathophysiology of diseases. Metabolomics technology examines low molecular weight substrates used in intracellular enzymatic reactions, intermediates and end products resulting from these reactions. Metabolomic examinations are gaining momentum in terms of understanding the pathophysiology of diseases, especially endometrial cancer and ovarian cancer, in the field of Obstetrics and Gynecology. Metabolomics continue to be investigated in understanding the pathophysiology of PCOS, but there are not enough studies yet on the effects of treatment on the disease in terms of metabolomics.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with polycystic ovary syndrome according to Rotterdam criteria and who do not have any additional chronic systemic disease

Exclusion Criteria:

* The presence of any diseases that cause hormonal disorders and any chronic systemic diseases, the patients who are already under any treatment for polycystic ovary syndrome

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-03 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Metabolomics | 3 months
  measured by H1 nuclear magnetic resonance spectroscopy

SECONDARY OUTCOMES:
hirsutism score | 3 months
  Measured by modified Ferriman Gallwey scoring system ranges between 0-36 points. Higher scores means worse outcome.
fasting serum insulin levels | 3 months
  measured on the 3rd day of menstrual cycle, before before 10 am, after 8-hour-night fasting. The lower levels means better outcome.
low density lipoprotein | 3 months
  measured on the 3rd day of menstrual cycle, before before 10 am, after 8-hour-night fasting. The lower levels means better outcome.
body mass index | 3 months
  weight and height will be combined to report BMI in kg/m^2. The lower index means better results.
clinical findings | 3 months
  Rising the number of participants with menstrual periods shorter than 35 days means better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes